CLINICAL TRIAL: NCT01566279
Title: A Two Parts, Biomarker Study to Identify Genetic Aberrations Predictive for Response on Everolimus in Solid Tumors Without Regular Treatment Options (CPCT-03)
Brief Title: A Study to Identify a Biomarker Predictive for Response on Everolimus in Solid Tumors (CPCT-03)
Acronym: CPCT-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, P.O. Witteveen, Investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL 37128.031.11; 2011-002562-20 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: solid tumors; all comers; everolimus; biomarker; next generation sequencing
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- everolimus (Other): All patients in first part will receive everolimus 10mg q.d.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — All patients will receive everolimus 10mg q.d.
  Other Names: Affinitor

SUMMARY:
The investigators hypothesize that certain mutations in the individual cancer genomes will predict response to Everolimus therapy. To identify possible genetic mutations that affect tumor response to Everolimus the investigators will obtain sequence analysis of tumors from all patients that will be treated with Everolimus in this study. Moreover, the investigators performed a systematic review of the currently available data to identify mutations that could be predictive for increased mTOR activity in cancer cells. These mutations have been described to lead to mTOR activation but their predictive value for response to Everolimus therapy remains unclear. The investigators will use the data generated in the investigators own prospective treatment study and the data from literature to select patients for entry into a second part of this trial. In this part the investigators want to test the hypothesis that selecting patients based on their specific genetic mutations increases the likelihood of response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up
* Inclusion in the CPCT-02 study
* Age ≥ 18 years
* Diagnosis of malignant tumor showing progressive disease according to investigators opinion
* WHO performance status of (0-2)
* Measurable disease allowing for volumetric measurements
* No availability of standard of care systemic treatment options or patient refuses to receive standard of care chemotherapy treatment
* A female is eligible to enter and participate in this study if she is of: Non-childbearing potential
* Adequate organ system function as defined in the protocol
* Fasting serum cholesterol ≤ 300 mg/dl or 7.75 mmol/L and fasting triglycerides ≤ 2.5 × ULN.

Exclusion Criteria:

* Previous treatment with mTOR inhibitors/pi3k inhibitors/AKT inhibitors
* Uncontrolled hypertension defined as RR > 160/95 mmHg
* Serious non-healing wound, ulcer or bone fracture
* Within 7 days of surgery (including minor procedures)
* Known and/or symptomatic intracerebral metastases
* Pregnancy or breast feeding, reproductive potential not using effective birth control methods
* Severe medical condition(s) prohibiting participation in the study
* Use of other investigational agents now or last 28 days prior to study treatment start
* Unable or unwilling to discontinue use of interacting medications or modify the dosing of interacting drugs for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study
* Less than four weeks after regular treatment/ palliative radiotherapy
* Prolongation of Fridericia corrected QT interval (QTcF) > 480 milliseconds
* Any severe and / or uncontrolled medical conditions such as:

  1. Unstable angina pectoris, symptomatic congestive heart failure myocardial infarction ≤6 months prior to enrollment, serious uncontrolled cardiac arrhythmia
  2. Uncontrolled diabetes as defined by fasting serum glucose > 1.5 × ULN
  3. Acute and chronic, active infectious disorders and nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy
  4. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs
  5. Significant symptomatic deterioration of lung function.
* Active, bleeding diathesis, or on oral anti-vitamin K medication (except low dose warfarin and acetylsalicylic acid or equivalent, as long as the INR is < 2.0)
* Patients with a known history of HIV seropositivity
* Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A within the last 5 days prior to enrollment
* Patients receiving concomitant immunosuppressive agents or chronic corticosteroids use, at the time of study entry except in cases outlined below:

  1. Topical applications (e.g. rash)
  2. Inhaled sprays (e.g. obstructive airways diseases),
  3. Eye drops
  4. Local injections (e.g. intra-articular) are allowed.
  5. Patients on stable low dose of corticosteroids for at least two weeks before enrollment are allowed in case of treatment of brain metastases .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
analyse a set of 1951 genes for prediction of response measured by time to progression (TTP) ratio (defined as the TTP without drug: TTP on drug) on mTOR inhibition. | An expected average of 5 months
  Inclusion until earliest date of disease progression (defined as a 30% volumetric increase in tumorvolume or appearance of new lesions)

SECONDARY OUTCOMES:
Progression free survival | An expected average of 4 months
  Time from initiation of everolimus to, either radiological (RECIST 1.1) or clinical disease progression or death from any cause.
Disease control rate (DCR) | At 3 months after initiation of everolimus
  Disease control rate (DCR) (DC = CR or PR or SD) as defined by RECIST 1.1 3 months after initiation of Everolimus.
Toxicity | An expected average of 6 months
  Toxicity will be assessed according to the Common Toxicity Criteria for Adverse Events (CTCAE) version v4.03: June 14, 2010
Median overall survival | An expected average of one year
  The (median) time from initiation of Everolimus to time of death or censored at the date of last follow-up. First analysis of overall survival will be performed within one year after inclusion of last subject.

CONTACTS AND LOCATIONS:
Overall Officials: M.H.G. Langenberg, MD/PhD, Principal Investigator — UMC Utrecht; N. Steeghs, MD/PhD, Principal Investigator — NKI-AvL; M.J.A. de Jonge, MD/PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - NKI-AVL, Amsterdam, North Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Cirkel GA, Weeber F, Bins S, Gadellaa-van Hooijdonk CG, van Werkhoven E, Willems SM, van Stralen M, Veldhuis WB, Ubink I, Steeghs N, de Jonge MJ, Langenberg MH, Schellens JH, Sleijfer S, Lolkema MP, Voest EE. The time to progression ratio: a new individualized volumetric parameter for the early detection of clinical benefit of targeted therapies. Ann Oncol. 2016 Aug;27(8):1638-43. doi: 10.1093/annonc/mdw223. Epub 2016 May 27. PMID 27234642
- See also: Related Info — http://www.cpct.nl